CLINICAL TRIAL: NCT00635895
Title: Comparison of Manual Lymph Drainage Therapy and Connective Tissue Massage in Females With Fibromyalgia: A Randomized Controlled Trial
Brief Title: Comparison of Lymph Drainage and Connective Tissue Massage in Fibromyalgia Patients
Acronym: FM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Collaborators: Hacettepe University (Other); Abant Izzet Baysal University (Other)
Responsible Party: Gamze Ekici, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Ekici - 3; ISRCTN12345678
Record Dates: First submitted 2008-03-06; First posted 2008-03-14 (Estimated); Last update posted 2008-03-14 (Estimated); Status verified 2008-03

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Manual Lymphatic Drainage; Connective Tissue Massage; Pain; Health Related Quality of Life; Randomized Controlled Trial
MeSH Terms: conditions — Fibromyalgia; Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Manual Lymph Drainage Therapy is a manual therapy method
  Interventions: Other: Manual Lymph Drainage Therapy and Connective Tissue Massage
- 2 (Active Comparator): Connective Tissue Massage
  Interventions: Other: Manual Lymph Drainage Therapy and Connective Tissue Massage

INTERVENTIONS:
Other: Manual Lymph Drainage Therapy and Connective Tissue Massage — The treatment program was carried out five times a week, during a 3-week period for both Manual Lymph Drainage Therapy and Connective Tissue Massage groups
  Other Names: No drug was used

SUMMARY:
The present study was designed to analyze and compare the effects of Manual Lymph Drainage Therapy and Connective Tissue Massage in females with Fibromyalgia (FM).

DETAILED DESCRIPTION:
The lack of specific disease mechanisms is reflected in the fact that no cure has been found for the disease. Thus, the many interventions which are advocated in FM are targeted against the more general characteristics of pain and disability. Current pharmacological interventions have limited efficacy. There is an increasing consensus that therapy should also include non-pharmacological approaches. Manual therapy techniques are composed of a variety of procedures directed at the musculoskeletal structures in the treatment of pain. Two major subcategories exist that divide these techniques into those which produce joint motion and those which do not. The first subcategory includes manipulation, mobilization, and manual traction. The second subcategory involves both generalized soft tissue therapies, such as the many types of massage, and focal soft tissue therapy (10).

Consequently, there is currently no recognized effective treatment for FM patients. In addition, there is limited number of study dealing with the effect of manual therapy techniques on FM. Although, there were some studies about Manual Lymph Drainage Therapy (MLDT) and Connective Tissue Massage (CTM) in FM. There wasn't found any study concerning the comparison of the effects of MLDT and CTM. In this study, MLDT and CTM were used for FM, which are included in the second subcategory of manual therapy techniques.

Based on positive results of some studies about MLDT and CTM in FM, this study was planned to test and compare the effects of MLDT and CTM in terms of pain, health status and HRQoL in females with FM using a randomized control trial.

ELIGIBILITY:
Inclusion Criteria:

* female outpatients
* being ≥ 25 years or older
* being met the criteria for FM as defined by the American College of Rheumatology
* having pain with the onset at least 3 months before baseline visit
* pain in the neck or shoulder region
* have never been treated for FM
* being volunteer for participating

Exclusion Criteria:

* pain from traumatic injury or structural or regional rheumatic disease,
* chronic infection,
* fever or an increased tendency to bleed,
* severe physical impairment,
* signs of tendinitis,
* cardiopulmonary disorder,
* inflammatory arthritis,
* autoimmune disease,
* uncontrolled endocrine disorder,
* allergic disorder,
* pregnancy or breast-feeding,
* malignancy,
* unstable medical or psychiatric illness or medication usage.
* They were asked not to use antidepressant, myorelaxant, and non-steroid anti-inflammatory drugs during three days before the first appointment and the treatment sessions and the evaluation process after the treatment.

Ages: 25 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2006-06; Primary Completion 2007-09 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Pain intensity VAS | 1 minute

SECONDARY OUTCOMES:
Fibromyalgia Impact Questionnaire (FIQ) | 10 minutes
algometry | 1 munute
Nottingham Health Profile | 10 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Gamze Ekici, PhD, Principal Investigator — Pamukkale University; Yesim Bakar, Asist. Prof., Study Director — Abant Izzet Baysal University; Turkan Akbayrak, Assoc.Prof., Study Director — Hacettepe University; Inci Yuksel, Prof, Study Director — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)